CLINICAL TRIAL: NCT01507402
Title: A Study to Assess the Safety and Tolerability of Single Ascending Doses of REGN1033(SAR391786)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R1033-HV-1107
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Cohort 1 (Experimental): Dose regimen 1 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 2 (Experimental): Dose regimen 2 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 3 (Experimental): Dose regimen 3 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 4 (Experimental): Dose regimen 4 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 5 (Experimental): Dose regimen 5 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 6 (Experimental): Dose regimen 6 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 7 (Experimental): Dose regimen 7 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 8 (Experimental): Dose regimen 3 (Participants > 65 to ≤ 85 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo
- Cohort 9 (Experimental): Dose regimen 9 (Participants 18 to ≤ 65 yrs old)
  Interventions: Drug: REGN1033(SAR391786); Drug: Placebo

INTERVENTIONS:
Drug: REGN1033(SAR391786) — Administration method A
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 8; Cohort 9
Drug: REGN1033(SAR391786) — Administration method B
  Arms: Cohort 5; Cohort 6; Cohort 7
Drug: Placebo — (inactive substance)

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose study to assess the safety and tolerability of Intravenous (IV) and Subcutaneous (SC) REGN1033(SAR391786) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and postmenopausal or surgically sterile females
2. Body mass index (BMI) between 18 and 30 kg/m2 inclusive
3. Willing and able to return for all clinic visits and complete all study-related procedures
4. Able to read and understand, and willing to sign the ICF

Exclusion Criteria:

1. Significant concomitant illness or history of significant illness such as, but not limited to cardiac, renal, rheumatologic, neurologic, psychiatric, endocrine, metabolic or lymphatic disease that would adversely affect the subject's participation in this study
2. History of muscle neoplasms such as rhabdomyoma, rhabdomyosarcoma, leiomyoma, leiomyosarcoma or uterine fibroid tumors
3. History of muscular dystrophy, myositis, and other primary diseases of skeletal muscle
4. History of heart diseases including but not limited to coronary heart disease with/without history of myocardial infarction, chronic or acute heart failure, or cardiac arrhythmia, valvular heart disease or cardiac hypertrophy. Subjects taking prophylactic aspirin are excluded from the study and should not discontinue taking prophylactic aspirin to participate in the study
5. History of systemic hypertension or use of concomitant medications to treat hypertension, or history of pulmonary hypertension
6. History of diabetes mellitus or gestational diabetes or use of concomitant medications for treatment of these
7. Recent use of androgenic steroids
8. Unexplained creatine phosphokinase (CPK) levels >3X upper limit of normal.
9. Any medical or psychiatric condition which, in the opinion of the investigator, would place the subject at risk, interfere with participation in the study or interfere with the interpretation of the study results
10. Women of childbearing potential (not surgically sterile or amenorrheic for at least twelve months if postmenopausal)
11. Onset of a new exercise routine or major change to a previous exercise or diet routine within 4 weeks prior to screening. Subjects must be willing to maintain his/her previous level of exercise for the duration of the study
12. Known history of seropositivity to human immunodeficiency virus (HIV) antibody; hepatitis B surface antigen or hepatitis C antibody (HCV) associated with a positive HCV RNA polymerase chain reaction at the screening visit
13. Positive urine drug test results during screening or history of drug or alcohol abuse within a year prior to the screening visit
14. Any hospitalization within 60 days prior to the screening visit
15. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives, whichever is longer, of the investigational drug, prior to the screening visit
16. History of a hypersensitivity reaction to doxycycline or to other tetracycline drugs
17. Previous exposure to any biological therapeutic agent, excepting vaccines

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of TEAEs | Day 1 to Day 113
  The primary endpoint in the study is the incidence and severity of TEAEs (Treatment Emergent Adverse Events) in subjects treated with REGN1033 or placebo, reported from the time of administration of study drug on day 1 (baseline) to completion of the study (day 113).

SECONDARY OUTCOMES:
Serum concentration | Baseline to End of Study (Day 113)
  To characterize the pharmacokinetic (PK) profile (i.e. serum concentration) of IV and SC doses of REGN1033.
Immunogenicity | Baseline to End of Study (Day 113)
  To assess the potential for immunogenicity following IV and SC doses of REGN1033.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Honolulu, Hawaii
  - Evansville, Indiana